CLINICAL TRIAL: NCT03581110
Title: CODP Imaging From a Dose Perspective - Effective Organ Doses of a Combined Inspiration-expiration Protocol on a 3rd Generation Dual-source CT
Brief Title: CODP Imaging From a Dose Perspective
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Joshua Gawlitza, Head of COPD imaging research, Universitätsmedizin Mannheim
Other Study IDs: UMannheim
Record Dates: First submitted 2018-06-22; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Radiation
Keywords: COPD; Computed tomography; Expiration; organ specific radiation dose
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Death | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- 16-slice CT scanner: 1426 patients that have received a noncontrast-enhanced chest CT on our 16-slice clinical routine CT scanner in inspiration only.
  Interventions: Diagnostic Test: computed tomography
- 2nd generation dual-source CT: 320 patients that have received a noncontrast-enhanced chest CT on our second generation dual-source CT scanner in inspiration only.
  Interventions: Diagnostic Test: computed tomography
- 3rd generation dual-source CT: 211 patients that have received a noncontrast-enhanced chest CT on our third generation dual-source CT scanner in inspiration and expiration.
  Interventions: Diagnostic Test: computed tomography

INTERVENTIONS:
Diagnostic Test: computed tomography — noncontrast-enhanced chest computed tomography

SUMMARY:
The noncontrast-enhanced chest computed tomography (CT) is an emerging diagnostical tool in patient with chronic obstructive pulmonary disease (COPD). As shown in previous studies and pointed out by the Fleischner society, an additional scan in expiration reflects the pathophysiology of this complex disease better and extends the clinical information of the CT.

Nevertheless, this scan is leading to an increase in radiation dose. But currently it is unclear if this increased radiation dose is proportional to the additional clinical value when compared to inspiration-only protocols. Therefore, the aim of this study was to compare the organ specific radiation doses of a combined inspiration-expiration CT on a 3rd generation dual-source scanner with noncontrast-enhanced chest CTs of two clinical routine scanners. Therefore, the radiation doses of nearly 2000 chest CTs have been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* noncontrast-enhanced chest CT performed on one of the named devices
* imaging performed between August 2014 and September 2017
* CT protocol used as previously specified

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The data was acquired retrospectively, by analyzing CT scans performed between August 2014 and September 2017. Further, the three different study groups have retrospectively been matched using the water equivalent diameter (WED). A difference of 5% was desired to eliminate a size related bias in the effective organ dose calculation.
Sampling Method: Non-Probability Sample
Enrollment: 1957 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
organ specific radiation doses | The organ dose calculations have been performed retrospectively. Therefore, the time frame is variable. The time set for the final outcome calculations was September 2017. Therefore, the time frame varies between 3 years and 1 week.
  Organ specific radiation doses of 17 individual organs

CONTACTS AND LOCATIONS:
Overall Officials: Joshua FM Gawlitza, MD, Principal Investigator — University medical center Mannheim; Holger Haubenreisser, MD, Principal Investigator — University medical center Mannheim; Frederik Trinkmann, MD, Principal Investigator — University medical center Mannheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coxson HO, Dirksen A, Edwards LD, Yates JC, Agusti A, Bakke P, Calverley PM, Celli B, Crim C, Duvoix A, Fauerbach PN, Lomas DA, Macnee W, Mayer RJ, Miller BE, Muller NL, Rennard SI, Silverman EK, Tal-Singer R, Wouters EF, Vestbo J; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Investigators. The presence and progression of emphysema in COPD as determined by CT scanning and biomarker expression: a prospective analysis from the ECLIPSE study. Lancet Respir Med. 2013 Apr;1(2):129-36. doi: 10.1016/S2213-2600(13)70006-7. Epub 2013 Feb 1. PMID 24429093
- [Background] Gawlitza J, Trinkmann F, Scheffel H, Fischer A, Nance JW, Henzler C, Vogler N, Saur J, Akin I, Borggrefe M, Schoenberg SO, Henzler T. Time to Exhale: Additional Value of Expiratory Chest CT in Chronic Obstructive Pulmonary Disease. Can Respir J. 2018 Mar 4;2018:9493504. doi: 10.1155/2018/9493504. eCollection 2018. PMID 29686742
- [Background] Haubenreisser H, Meyer M, Sudarski S, Allmendinger T, Schoenberg SO, Henzler T. Unenhanced third-generation dual-source chest CT using a tin filter for spectral shaping at 100kVp. Eur J Radiol. 2015 Aug;84(8):1608-1613. doi: 10.1016/j.ejrad.2015.04.018. Epub 2015 Apr 28. PMID 26001437
- [Background] Gordic S, Morsbach F, Schmidt B, Allmendinger T, Flohr T, Husarik D, Baumueller S, Raupach R, Stolzmann P, Leschka S, Frauenfelder T, Alkadhi H. Ultralow-dose chest computed tomography for pulmonary nodule detection: first performance evaluation of single energy scanning with spectral shaping. Invest Radiol. 2014 Jul;49(7):465-73. doi: 10.1097/RLI.0000000000000037. PMID 24598443
- [Background] Braun FM, Johnson TR, Sommer WH, Thierfelder KM, Meinel FG. Chest CT using spectral filtration: radiation dose, image quality, and spectrum of clinical utility. Eur Radiol. 2015 Jun;25(6):1598-606. doi: 10.1007/s00330-014-3559-1. Epub 2014 Dec 17. PMID 25515204